CLINICAL TRIAL: NCT03419585
Title: Systematic Light Exposure to Prevent Fatigue in Prostate Cancer Patients
Brief Title: The "PC-LIGHT" Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Lisa M. Wu, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00205260
Record Dates: First submitted 2018-01-24; First posted 2018-02-05 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer; Sleep; Depression; Fatigue; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms; Depression; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized to one of two arms: an intervention light group or a comparison light group. Both the participant and the investigator will be blind to the light assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention light (Experimental): 30 minutes of intervention systematic light exposure daily for the course of radiation therapy (approximately 8 weeks).
  Interventions: Device: Intervention systematic light exposure
- Comparison light (Active Comparator): 30 minutes of comparison systematic light exposure daily for the course of radiation therapy (approximately 8 weeks).
  Interventions: Device: Comparison systematic light exposure

INTERVENTIONS:
Device: Intervention systematic light exposure — 30 minutes of intervention systematic light exposure daily
  Arms: Intervention light
Device: Comparison systematic light exposure — 30 minutes of comparison systematic light exposure daily
  Arms: Comparison light

SUMMARY:
Fatigue due to cancer and its treatment (for example, radiation therapy) can interfere with quality of life and can linger long after treatment has ended, yet research examining preventative approaches has produced limited clinical benefit. The proposed study will provide information about systematic light exposure for the prevention of fatigue in prostate cancer patients undergoing radiation therapy and will investigate how it works. This study would facilitate the development of this potential preventative treatment, giving health care providers and cancer survivors a much-needed tool to help with cancer-related fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with clinical localized prostate cancer,
* Are about to begin external beam radiation therapy (RT) for prostate cancer,
* Are 18 years of age or older,
* Are able to speak or read English,
* Have internet access.

Exclusion Criteria:

* History of light therapy use (e.g. systematic light exposure),
* Active infection
* History of chronic fatigue disorders
* Confounding underlying medical illnesses such as significant pre-existing anemia (Hb<10 gm/dl)
* Diagnosed or suspected psychiatric or medical condition that might contribute to fatigue (other than those caused by the cancer or its treatment)
* Hypothyroidism or documented history of hypothyroidism on thyroid replacement hormone within <3 months of initiating RT
* History of bipolar disorder or mania
* History of seasonal affective disorder
* Diagnosed sleep apnea, restless legs, or other sleep disorders (not including insomnia) known to affect fatigue
* Use of photosensitizing medication
* Plans to travel across more than 2 time zones during the study
* Shift worker
* Adults unable to consent, individuals who are not yet adults, pregnant women, and prisoners will be excluded from the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Fatigue FACIT-Fatigue scores | Baseline
  FACIT-Fatigue scores
Fatigue | Change from Baseline to the 4th week of the intervention
  FACIT-Fatigue scores
Fatigue | Change from Baseline to the 8th week of the intervention
  FACIT-Fatigue scores
Fatigue | Change from Baseline to 2 months after the intervention
  FACIT-Fatigue scores

SECONDARY OUTCOMES:
Circadian activity rhythms | Baseline
  Actigraphy
Circadian activity rhythms | During the 4th week of the intervention
  Actigraphy
Circadian activity rhythms | During the 8th week of the intervention
  Actigraphy
Circadian activity rhythms | 2 months after the intervention
  Actigraphy
Sleep quality | Baseline
  Pittsburgh Sleep Quality Index (PSQI)
Sleep quality | During the 4th week of the intervention
  Pittsburgh Sleep Quality Index (PSQI)
Sleep quality | During the 8th week of the intervention
  Pittsburgh Sleep Quality Index (PSQI)
Sleep quality | 2 months after the intervention
  Pittsburgh Sleep Quality Index (PSQI)
Depressed mood | Baseline
  Center for Epidemiologic Studies Depression Scale (CESD). Score range is 0 to 60, where higher scores represent more symptomatology present.
Depressed mood | During the 4th week of the intervention
  Center for Epidemiologic Studies Depression Scale (CESD). Score range is 0 to 60, where higher scores represent more symptomatology present.
Depressed mood | During the 8th week of the intervention
  Center for Epidemiologic Studies Depression Scale (CESD). Score range is 0 to 60, where higher scores represent more symptomatology present.
Depressed mood | 2 months after the intervention
  Center for Epidemiologic Studies Depression Scale (CESD). Score range is 0 to 60, where higher scores represent more symptomatology present.
Cognitive Functioning | Baseline
  Psychometric Analysis of the Patient Assessment of Own Functioning Inventory (PAOFI)
Cognitive Functioning | During the 4th week of the intervention
  Psychometric Analysis of the Patient Assessment of Own Functioning Inventory (PAOFI)
Cognitive Functioning | During the 8th week of the intervention
  Psychometric Analysis of the Patient Assessment of Own Functioning Inventory (PAOFI)
Cognitive Functioning | 2 months after the intervention
  Psychometric Analysis of the Patient Assessment of Own Functioning Inventory (PAOFI)
Sexual and urinary functioning | Baseline
  3 items from the Sexual Adjustment Questionnaire & 3 items from American Urological Association (AUA) symptom index
Sexual and urinary functioning | During the 4th week of the intervention
  3 items from the Sexual Adjustment Questionnaire & 3 items from American Urological Association (AUA) symptom index
Sexual and urinary functioning | During the 8th week of the intervention
  3 items from the Sexual Adjustment Questionnaire & 3 items from American Urological Association (AUA) symptom index
Sexual and urinary functioning | 2 months after the intervention
  3 items from the Sexual Adjustment Questionnaire & 3 items from American Urological Association (AUA) symptom index
Cognitive functioning | Baseline
  Neuropsychological tests
Cognitive functioning | During the 8th week of the intervention
  Neuropsychological tests
Cognitive functioning | 2 months after the intervention
  Neuropsychological tests
Health-related quality of life | Baseline
  Functional Assessment of Cancer Therapy - Prostate (FACT-P). From Radiation Therapy Oncology Group: "The FACT-P is a multidimensional, self-report QoL instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being."with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being.
Health-related quality of life | During the 4th week of the intervention
  Functional Assessment of Cancer Therapy - Prostate (FACT-P). From Radiation Therapy Oncology Group: "The FACT-P is a multidimensional, self-report QoL instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being."
Health-related quality of life | During the 8th week of the intervention
  Functional Assessment of Cancer Therapy - Prostate (FACT-P). From Radiation Therapy Oncology Group: "The FACT-P is a multidimensional, self-report QoL instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being."with prostate cancer patients (1, 2, 3). It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being.
Health-related quality of life | 2 months after the intervention
  Functional Assessment of Cancer Therapy - Prostate (FACT-P). From Radiation Therapy Oncology Group: "The FACT-P is a multidimensional, self-report QoL instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being."with prostate cancer patients (1, 2, 3). It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being.

OTHER OUTCOMES:
Credibility/Expectancy | Baseline
  Credibility/Expectancy questionnaire. There are two scales used during the questionnaire - (1-9, and 0-100%). A composite score can be calculated for each factor (expectancy and credibility).
Treatment satisfaction | During the 8th week of the intervention
  Functional Assessment of Cancer Therapy - Treatment Satisfaction - General (FACT-TS-G)
Usage of light box | Throughout intervention period (8 weeks)
  integrated meter measurement and Litebook log. Length of time light box has been used.
Chronotype | Baseline
  Morningness-eveningness questionnaire. From the item itself: "Scores can range from 4-25. Scores of 7 and below indicate "evening types." Scores of 22 and above indicate "morning types." Scores between 8-21 indicate "intermediate types."
BMI | Baseline
  BMI table
Physical health | Baseline
  Goldin Leisure Time Exercise Questionnaire. From the measure itself: " For the first question, weekly frequencies of strenuous, moderate, and light activities are multiplied by nine, five, and three, respectively. Total weekly leisure activity is calculated in arbitrary units by summing the products of the separate components, as shown in the following formula: Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light) The second question is used to calculate the frequency of weekly leisure-time activities pursued "long enough to work up a sweat" (see questionnaire)."

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Wu, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Univeristy Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No